CLINICAL TRIAL: NCT06781593
Title: Effects of Light Therapy on Compliance With Continuous Positive Airway Pressure in a Population of Depressed Patients Newly Fitted With Devices for Obstructive Sleep Apnea
Brief Title: Combining Light Therapy and CPAP in Depression
Acronym: LUCIOPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-A01551-46
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depression; Sleep Architecture; Obstructive Sleep Apnea; Compliance; Continuous Positive Airway Pressure (CPAP); Light Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Apnea, Obstructive; Patient Compliance | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized sham controlled clinical trial, single center, double-blind, parallel group-controlled two arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sham light therapy consists of using a device similar to the active condition (glasses) but delivering a weakened version of the active light (addition of a filter and reduction of light intensity), emitting an intensity of 33 lux and a light spectrum (600 nm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Light therapy (Active Comparator): Active light therapy comes in the form of glasses and emits an intensity of 1200 Lux and a cyan-colored light spectrum (500nm), corresponding to a retinal exposure of 361.91uW/cm2 with a 30-min daily exposure upon waking for 2 weeks
  Interventions: Device: Light therapy
- Sham Light therapy (Placebo Comparator): Sham light therapy is the same device but in an attenuated version (addition of a filter and reduction of light intensity), emitting an intensity of 33 Lux and a light spectrum (600 nm) with a 30-min daily exposure upon waking for 2 weeks.
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — The intervention consists of 30 minutes of daily exposure to light therapy glasses (active or sham according to randomization) on waking for 2 weeks. The light therapy will be delivered in the patient's home at the same time as CPAP is introduced.

SUMMARY:
In a double-blind, parallel-group controlled trial, we aim to measure the effect of two weeks of light therapy combined with the CPAP on compliance CPAP in patients with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a frequent and disabling psychiatric condition. Clinically, MDD is characterized by persistent depressed mood, loss of interest, loss of pleasure in daily activities, and sleep disturbance. The link between sleep disturbance and depressive symptoms is complex and bidirectional, but data from the literature suggest that treatment of sleep disturbance in patients with MDD is associated with a better prognosis and a reduction in the number of relapses.

Among sleep disorders, obstructive sleep apnea syndrome (OSAS) is a frequent comorbidity in MDD. The severity of OSAS correlates with the severity of depressive symptoms, and treatment of OSAS with continuous positive airway pressure (CPAP) can reduce daytime sleepiness and some depressive symptoms. Despite its efficacy, CPAP treatment is often poorly tolerated by patients, and compliance rates are often low, with discontinuation of treatment within the first 15 days of initiation, before it has had a chance to demonstrate its effectiveness. Light therapy is a non-invasive medical device that has been shown to rapidly reduce certain depressive symptoms, such as insomnia.

The aim of the study is to investigate whether the combination of two weeks of active light therapy with the introduction of CPAP can increase CPAP compliance at two weeks of treatment (D14) in patients with MDD and OSAS.

To this end, 130 patients with MDD (MADRS > 15) will be recruited and randomized to two intervention groups: one group receiving active light therapy combined with CPAP and one group receiving sham light therapy combined with CPAP. The study will take place in the patient's home. The company's service providers, accustomed to installing CPAP in patients' homes, will be responsible for delivering the light therapy glasses and actimetry watches at the end of the 2-week treatment period. A polysomnography recording will be acquired prior to treatment. Quality and compliance measurements are recorded by the CPAP machines and will be statistically analyzed.

The investigators hypothesize that the early combination of active light therapy and CPAP will enable changes in CPAP complance, MDD symptoms severity, and sleep quality in patients with MDD and OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Adults consulting at the MICHEL JOUVET unit, CH Le Vinatier, Bron
* Adults with a diagnosis of major depressive episode (DSM-V) and with a MADRS score ≥ 15
* Adults with a diagnosis of OSAS on ventilatory polygraphy or polysomnography (AASM 2017 criteria) requiring CPAP.

Exclusion Criteria:

* Refusal to participate.
* Pregnant and breast-feeding women
* Under guardianship or curatorship.
* Unstable psychiatric or physical pathology (e.g., hypomania, high suicidal risk) considered incompatible with the study by the investigators.
* Other psychiatric, neurologic or somatic conditions
* Contraindication to light therapy: retinopathy, retinitis pigmentosa, diabetic retinopathy, macular degeneration, glaucoma, recent eye surgery (less than 3 months).

patient wishing to choose a provider other than the protocol provider.

* Patient wishing to choose a device other than SEFAM's S-BOX or a mask other than the nasal mask at the time of introduction.
* Nasal obstruction.
* Refusal to use actimetry, refusal to use light therapy, refusal to use CPAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
CPAP Compliance | 1 time :Day 14
  CPAP compliance will be measured via CPAP reports on manufacturers' websites. Analysis of time spent with CPAP per night of sleep (with a cut off score set at 4 hours or more per night = compliant patient)

SECONDARY OUTCOMES:
The maintenance of the effect ot the intervention will be measured 14 days before the interruption of light therapy at D28 | 3 times :The MADRS score will be measured during the inclusion visit (Day 7) and at Day 28, 14 days after the stop of light therapy
  MADRS, is a standardized clinical scale used to assess the severity of depression in patients with mood disorders (score from 0 to over 34 = from healthy to severe depression). This hetero-questionnaire will be completed by a trained psychiatrisy during the inclusion visit and after the intervertion (D28). Analysis of the variation in the MADRS score makes it possible to determine the effect of light therapy on the evolution of the patient's depressive state.
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - ISI (Insomnia Severity Index): 0-7 (No insomnia), 8-14 (Sub-clinical insomnia), 15-21 (Clinical insomnia (moderate)), 22-28 (Clinical insomnia (severe))
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - PSQI (Pittsburgh Sleep Quality Index). Score has a possible range of 0-21 points. Actual scores ranged from 0 to 20 points, with an overall group mean of 7.4, median of 6.0, and SD of 5.1.
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - PFS (Pichot Fatigue Scale): A total of more than 22, out of a maximum of 32, indicates excessive fatigue which should be investigated.
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - ESS (Epworth Sleepiness Scale): 0-5 (lower normal daytime sleepiness), 6-10 (normal daytime sleepiness), 11-12 (mild excessive daytime symptoms), 13-15 (moderate excessive daytime symptoms), 16-24 (severe excessive daytime symptom).
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - Beck (BDI-13): 0-4 (no depression), 4-7 (mild depression), 8-15 (moderate depression), 16 and over (severe depression)
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - HAD (Hospital Anxiety Depression Scale) anxiety section: 7 or less (no symptomatology), 8 to 10 (doubtful symptomatology), 11 and more (definite symptomatology)
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - Mac Nair Memory Complaint Scale (39 items rated from 0 to 4, i.e. from 0 to 156)
self-questionnaires form | 3 times :Several self-questionnaires will be completed three times: at inclusion (Day 0), after 14 days (removal of light therapy glasses; Day 14) and at end-point (Day 28)
  - MCTQ (Munich Chronotype) Total scores can range from 16 to 86, with the lowest values representing extreme-late chronotypes.
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Total sleep time in minutes.
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Sleep onset delay (in minutes).
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Time in bed in minutes.
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Sleep efficiency in percentage (TST on TPL)
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Sleep fragmentation in minutes (intra-sleep wake duration).
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Sleep onset latency.
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Motor activity in absolute value.
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Daily nap time in minutes.
Actimetry results | 3 times :average of different parameters over the periods before inclusion, from Day 7 to Day 0 (base line), period of treatment from Day 0 to Day 14 (CPAP and light therapy), period of CPAP without light therapy from Day14 to Day 28 (CPAP alone)
  Average of the following parameters over the different periods :
  - Light exposure in lux.
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Delay in onset of REM sleep (in minutes).
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Amount of REM sleep (SP in minutes).
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Amount of deep slow wave sleep (SLP in minutes).
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Ratio (SLP + SP) / TST.
polysomnography results, sleep architecture | 2 times :baseline measure to control for OSAS diagnosis (performed between Day 30 and Day 1), and after intervention measure (post-PPC + light therapy at Day 28)
  Average of the following parameters over the different periods
  - Arousal/microarousal index per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien S CATOIRE, DR, Principal Investigator — Centre Hospitalier le Vinatier
Locations (2):
- France (2):
  - Centre Hospitalier le Vinatier, Bron, France
  - Centre Hospitalier le Vinatier, Bron

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Azzaoui H, Catoire S, Lecharpentier H, Felician J, Grasset O, Gronfier C, Vallet W, D'amato T, Brunelin J. Adjunctive bright light therapy to enhance continuous positive airway pressure adherence in patients with comorbid major depressive disorder and obstructive sleep apnoea syndrome: study protocol for a randomised sham-controlled trial. BMJ Open. 2025 Dec 15;15(12):e108669. doi: 10.1136/bmjopen-2025-108669. PMID 41401997